CLINICAL TRIAL: NCT02550457
Title: Effects of Kinesio Taping on Chronic Nonspecific Low Back Pain: a Randomized Controlled Trial
Brief Title: Kinesio Taping on Chronic Nonspecific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Jamilson Simões Brasileiro, Professor of Physiotherapy, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 056666/2015
Record Dates: First submitted 2015-09-11; First posted 2015-09-15 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control group (No Intervention): It will not apply any tape.
- Experimental group 1 (Experimental): Apply the KT with tension in the erector spine muscles.
  Interventions: Other: Functional elastic tape tensioned
- Experimental group 2 (Experimental): Apply the KT without tension in the erector spine muscles.
  Interventions: Other: Functional elastic tape non-tensioned
- Placebo group (Placebo Comparator): Apply Micropore tape in the erector spine muscles.
  Interventions: Other: Rigid Tape

INTERVENTIONS:
Other: Functional elastic tape tensioned — Application of Kinesio Taping with tension in the erector spine muscles.
  Other Names: Kinesio Taping with tension
  Arms: Experimental group 1
Other: Functional elastic tape non-tensioned — Application of Kinesio Taping without tension in the erector spine muscles.
  Other Names: Kinesio Taping without tension
  Arms: Experimental group 2
Other: Rigid Tape — Application of Micropore tape in the erector spine muscles.
  Other Names: Micropore Tape
  Arms: Placebo group

SUMMARY:
This study propose analyze the effects of Kinesio Taping® in chronic nonspecific low back pain. All the subjects will be submitted to an evaluation of the painful sensation, functional performance, trunk range of motion and neuromuscular performance at three different times.

ELIGIBILITY:
Inclusion Criteria:

* Female between 18 and 50 years of age with chronic nonspecific low back pain for more than three months.

Exclusion Criteria:

* Serious spinal pathologies (fractures, tumors, and inflammatory pathologies such as ankylosing spondylitis);
* Nerve root compromise (disc herniation and spondylolisthesis with neurological compromise, spinal stenosis, and others);
* Fibromyalgia
* Corticosteroid treatment in the previous two weeks;
* Antiinflammatory treatment in the previous 24 hours;
* Contraindications to the use of Kinesio Taping (allergy or intolerance);
* Score of two or less on Visual Analogue Scale of the first day;
* Pregnancy;
* Previous Kinesio Tape therapy on lumbar.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2015-09; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Painful sensation | Evaluation of pain sensation three days after the application of the tape.
  Pain sensation measured by pain numerical rating scale

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal do Rio Grande do Norte, Natal, Rio Grande do Norte, Brazil

REFERENCES:
- [Derived] Macedo LB, Richards J, Borges DT, Melo SA, Brasileiro JS. Kinesio Taping reduces pain and improves disability in low back pain patients: a randomised controlled trial. Physiotherapy. 2019 Mar;105(1):65-75. doi: 10.1016/j.physio.2018.07.005. Epub 2018 Jul 26. PMID 30348455